CLINICAL TRIAL: NCT00375726
Title: Phase 1 Study of the Safety and Immunogenicity of rDEN3/4delta30(ME), a Live Attenuated Virus Vaccine Candidate for the Prevention of Dengue Serotype 3
Brief Title: Safety of and Immune Response to a Dengue Virus Vaccine (rDEN3/4delta30[ME]) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Anna Durbin, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 228; WIRB Protocol Number 20061667
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Dengue
Keywords: Dengue Fever; Dengue Vaccine; Dengue Virus; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): One subcutaneous vaccination with rDEN3/4delta30(ME) vaccine (10^3 PFU dose) into the deltoid region of either arm.
  Interventions: Biological: rDEN3/4delta30(ME)
- 2 (Experimental): One subcutaneous vaccination with rDEN3/4delta30(ME) vaccine (10^5 PFU dose) into the deltoid region of either arm. This arm may enroll after Arm 1 depending on the immunological response of Arm 1.
  Interventions: Biological: rDEN3/4delta30(ME)
- 3 (Experimental): One subcutaneous vaccination with rDEN3/4delta30(ME) vaccine (10^1 PFU dose) into the deltoid region of either arm. This arm may enroll after Arm 1 depending on the immunological response of Arm 1.
  Interventions: Biological: rDEN3/4delta30(ME)
- 4 (Placebo Comparator): One subcutaneous vaccination with placebo into the deltoid region of either arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rDEN3/4delta30(ME) — Live attenuated rDEN3/4delta30(ME) vaccine (one of three doses)
  Arms: 1; 2; 3
Biological: Placebo — Placebo for rDEN3/4delta30(ME)
  Arms: 4

SUMMARY:
Dengue fever, caused by dengue viruses, is a major health problem in the tropical and subtropical regions of the world. The purpose of this study is to test the safety of and immune response to a new dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses, which cause dengue fever and dengue shock syndrome, are a major cause of morbidity and mortality in several of the world's tropical and subtropical regions. The rDEN3/4delta30(ME) vaccine is a live attenuated dengue virus vaccine that may be protective against dengue virus serotype 3 (DEN3). The purpose of this study is to evaluate the safety and immunogenicity of the rDEN3/4delta30(ME) vaccine in healthy adults.

This study will last 40 weeks. Participants will be randomly assigned to receive one of three doses of rDEN3/4delta30(ME) or placebo. Participants in Group 1 will receive the middle dose of rDEN3/4delta30(ME) or placebo at study entry. Group 2a will begin enrollment after the immunogenicity review of all participants in Group 1. Participants in Group 2a will receive the highest dose of rDEN4delta30(ME) or placebo at study entry. Group 2b will begin enrollment after the immunogenicity review of all participants in Group 2a. Participants in Group 2b will receive the lowest dose of rDEN4delta30(ME) or placebo.

After vaccination, participants in all groups will be followed closely every other day for the first 16 days of the study. Participants will take their temperature three times a day through Day 16 and record each measurement in a diary. After Day 16, participants will have study visits on Days 21, 28, 42, and 180; a physical exam and blood collection will occur at all visits. Some participants may be asked to join a skin biopsy substudy.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Available for the duration of the study
* Willing to use acceptable forms of contraception for the duration of the study

Exclusion Criteria:

* Significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, may interfere with the study
* Significant laboratory abnormalities
* Medical, work, or family problems as a result of alcohol or illegal drug use within 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Emergency room visit or hospitalization for severe asthma within 6 months prior to study entry
* HIV-1 infected
* Hepatitis C virus (HCV) infected
* Hepatitis B surface antigen positive
* Immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive medications within 30 days prior to study entry. Participants using topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Absence of spleen
* Blood products within 6 months prior to study entry
* Previous dengue virus or other flavivirus (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus) infection
* Previously received yellow fever or dengue vaccine
* Plans to travel to an area where dengue infection is common
* Received an investigational agent within 30 days prior to study entry
* Other condition that, in the opinion of the investigator, would interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety, as defined by frequency of vaccine-related adverse events, as classified by both intensity and severity through active and passive surveillance | Throughout study
Immunogenicity, as determined by anti-DEN3 neutralizing antibody measured on Days 0, 21, 28, 42, and 180 | Throughout study

SECONDARY OUTCOMES:
Assess the frequency, quantity, and duration of viremia in each dose cohort studied | Throughout study
Determine the number of vaccinees infected with rDEN3/4delta30(ME) | Throughout study
Determine cellular targets of vaccine infection, including peripheral blood mononuclear cells (PBMCs) and skin from participants who are willing to undergo skin biopsy | Throughout study
Compare the infectivity rates, safety, and immunogenicity between dose groups | At study completion
Evaluate the immunopathological mechanism of vaccine-associated rash in those volunteers who are willing to undergo skin biopsy | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, Johns Hopkins School of Public Health
Locations (1):
- Center for Immunization Research, Baltimore, Maryland, United States

REFERENCES:
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Development of a live attenuated dengue virus vaccine using reverse genetics. Viral Immunol. 2006 Spring;19(1):10-32. doi: 10.1089/vim.2006.19.10. PMID 16553547
- [Background] Blaney JE Jr, Hanson CT, Firestone CY, Hanley KA, Murphy BR, Whitehead SS. Genetically modified, live attenuated dengue virus type 3 vaccine candidates. Am J Trop Med Hyg. 2004 Dec;71(6):811-21. PMID 15642976
- [Background] Blaney JE Jr, Matro JM, Murphy BR, Whitehead SS. Recombinant, live-attenuated tetravalent dengue virus vaccine formulations induce a balanced, broad, and protective neutralizing antibody response against each of the four serotypes in rhesus monkeys. J Virol. 2005 May;79(9):5516-28. doi: 10.1128/JVI.79.9.5516-5528.2005. PMID 15827166
- [Background] Durbin AP, Whitehead SS, McArthur J, Perreault JR, Blaney JE Jr, Thumar B, Murphy BR, Karron RA. rDEN4delta30, a live attenuated dengue virus type 4 vaccine candidate, is safe, immunogenic, and highly infectious in healthy adult volunteers. J Infect Dis. 2005 Mar 1;191(5):710-8. doi: 10.1086/427780. Epub 2005 Jan 27. PMID 15688284